CLINICAL TRIAL: NCT01773005
Title: A Single Center, Randomized, Open-Label Trial to Compare the Safety and Efficacy of Caldolor Used Singly and in Combination With Ofirmev in Total Knee or Hip Arthroplasty Surgery Patients
Brief Title: Caldolor Versus Caldolor Plus OFIRMEV in Total Knee or Hip Arthroplasty Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anita Gupta (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Anita Gupta, Associate Professor, Hahnemann University Hospital
Organization: Hahnemann University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CP-001-12; 20121232 (Other Grant/Funding Number: Cumberland)
Record Dates: First submitted 2013-01-09; First posted 2013-01-21 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: Anesthetics, Intravenous
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caldolor (Sham Comparator): Subject receives the interventional drug, intravenous ibuprofen (800 mg Caldolor) at the induction of anesthesia, followed by 800 mg Caldolor every 6 hours until discharge or for a total of up to 120 hours (5 days)
  Interventions: Drug: Caldolor
- Ofirmev (Active Comparator): Subject receives the interventional drug, intravenous ibuprofen (800 mg Caldolor) at the induction of anesthesia and intravenous Acetaminophen (1000 mg Ofirmev) at the time of surgical wound closure, followed by 800 mg Caldolor plus 1000 mg Ofirmev every 6 hours until discharge for a total of up to 120 hours (5 days)
  Interventions: Drug: Ofirmev; Drug: Caldolor

INTERVENTIONS:
Drug: Ofirmev — Subject receives the interventional drug, intravenous ibuprofen (800 mg Caldolor) at the induction of anesthesia and intravenous Acetaminophen (1000 mg Ofirmev) at the time of surgical wound closure, followed by 800 mg Caldolor plus 1000 mg Ofirmev every 6 hours until discharge for a total of up to 120 hours (5 days)
  Other Names: Intravenous Acetaminophen
  Arms: Ofirmev
Drug: Caldolor — Subject receives the interventional drug, intravenous ibuprofen (800 mg Caldolor) at the induction of anesthesia, followed by 800 mg Caldolor every 6 hours until discharge or for a total of up to 120 hours (5 days)
  Other Names: Intravenous Ibuprofen

SUMMARY:
The objective of this study is to compare the effectiveness and of perioperative use of Caldolor alone and in combination with OFIRMEV in total knee or hip arthroplasty procedures.

DETAILED DESCRIPTION:
Patients undergoing total knee or hip arthroplasty procedures at University Pain Institute at Hahnemann will be included in this study.

Following Institutional Review Board's approval, eligible patients will be selected from the Pre Admission Testing for total knee or hip arthroplasty surgeries planned at Hahnemann University Hospital.

The cases will be randomized in a 1:1 ratio into either Group 1 or Group 2. Group 1 will receive 800 mg Caldolor at the induction of anesthesia, followed by 800 mg Caldolor every 6 hours until discharge or for a total up to 120 hours (5 days) Group 2 will receive 800 mg Caldolor at the induction of anesthesia and 1000 mg Ofirmev at the time of surgical wound closure, followed by 800 mg Caldolor plus 1000 mg Ofirmev every 6 hours until discharge or for a total up to 120 hours (5 days)

After the surgery, at the request of the patient they could receive morphine administered by patient-controlled analgesia pump, or by hospital staff.

The analgesics and procedures involved in this study are all standard of care drugs prescribed and administered by the attending anesthesiologist for control of total knee or hip arthroplasty surgery related pain. Data collected for every patient will exist in the patient's medical chart as part of their standard medical care. No additional patient procedures or activities are mandated by this study.

The data collection and analysis will be completed in duration of 1 year

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18-70 scheduled for total knee or hip arthroplasty surgery
* American Society of Anesthesiology physical status I, II, III

Exclusion Criteria:

* Impaired liver function
* History of substance abuse or chronic pain
* Patients known to be hypersensitive to any of the components of Caldolor or Ofirmev
* Patients less than 18 years of age.
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions.
* Be pregnant or nursing
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score (VAS) | Before surgery to Post-operative Day 5 (or Hospital Discharge)
  First Post-op 100mm VAS pain score at rest and with movement

SECONDARY OUTCOMES:
Quality of Recovery (QoR40 scale) | Post-operative Day one
  Patient satisfaction score

OTHER OUTCOMES:
Side effects | Post-operative Day one to five (or hospital discharge)
  Incidence of opioid-related side effects

CONTACTS AND LOCATIONS:
Overall Officials: Kirtanaa Voralu, MS, Study Director — Associate Director Research Management
Locations (1):
- University Pain Institute Hahnemann Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No